CLINICAL TRIAL: NCT05583955
Title: A Double-blind, Placebo-controlled, Phase IIb, Multi-center, Ten-week Prospective Study to Evaluate the Efficacy and Safety of NOE-105 in Adult Male Patients With Childhood Onset Fluency Disorder (Orpheus)
Brief Title: A 10-week Efficacy Study of NOE-105 in Childhood Onset Fluency Disorder (Orpheus)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noema Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOE-CFD-201
Record Dates: First submitted 2022-06-16; First posted 2022-10-18 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2024-03

CONDITIONS: Childhood-Onset Fluency Disorder
MeSH Terms: conditions — Childhood-Onset Fluency Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Escalating doses of NOE-105 capsules
  Interventions: Drug: NOE-105
- Placebo (Placebo Comparator): Escalating doses of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NOE-105 — Escalating dose levels of NOE-105 will be given and maximum tolerated dose will be maintained
  Other Names: Escalating dose levels of NOE-105
  Arms: Active
Drug: Placebo — Escalating dose levels of matching Placebo will be given
  Other Names: Placebo to match
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the effectiveness of NOE-105 on speech fluency without the known antipsychotic-induced side effects of commonly used treatments for childhood onset fluency disorder (COFD).

DETAILED DESCRIPTION:
NOE-105 is an investigational selective PDE10A inhibitor with a potential therapeutic effect for the treatment of COFD. In this study adult male patients may be randomized to a double-blind, placebo-controlled, parallel group treatment with NOE-105 or placebo once daily. The study is designed to find the maximum tolerated dose of NOE-105 and thereafter, to maintain the participants at this dose until they have completed a total of 10 weeks treatment period. Following up to 10 weeks of treatment, participants will visit the study site for a follow-up visit within 28 (± 7) days of the date of the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
2. Patients who satisfy DSM-5 criteria for childhood onset fluency disorder and are suitable for pharmacotherapy.
3. Have a history of stuttering for more than or equal to ≥ 2 years with onset consistent to developmental in nature before age 8 years.
4. Patient reported global stuttering experience as "moderate" at screening and baseline.
5. Patients must discontinue all medications used to treat stuttering for at least 14 days prior to receiving study treatment. With the exception of antipsychotic therapies (see exclusion criterion #11), other psychotropic drugs will be allowed provided they have been stable for at least 14 days prior to receiving study treatment and are expected to remain stable for the duration of the study.
6. BMI within the range 19 to 35 kg/m2 (inclusive).
7. Male Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male patients must use a condom during the treatment period and until the end of relevant systemic exposure in the male participant, plus a further 90-day period. In addition, for a non-pregnant WOCBP partner.
8. Capable of giving signed informed consent
9. Able to read and write in English

Exclusion Criteria:

1. Stuttering is related to a known neurological cause eg, stroke, etc.
2. Low IQ in the opinion of the investigator.
3. Patients with uncontrolled seizure disorders.
4. A history of severe traumatic brain injury or stroke.
5. Patients who are, in the investigator's opinion, at imminent risk of suicide.
6. Known to have tested positive for human immunodeficiency virus.
7. Known DSM-5 diagnosis of substance abuse or dependence.
8. Unstable medical illness or clinically significant abnormalities on screening tests/exams.
9. Any unstable medical conditions or are currently ill (eg, congenital heart disease, arrhythmia or cancer), which, in the investigator's judgment, will put them at a risk of major adverse event during this trial, are expected to progress during the study, or will interfere with safety and efficacy assessments.
10. Initiation of new behavioral therapies for stuttering within 10 weeks prior to baseline.
11. Use of antipsychotic drug therapy within 14 days prior to receiving treatment until the EoT visit.
12. Participation in another clinical study with an IP administered in the last 30 days.
13. Participants with a known hypersensitivity to NOE-105 or any of the excipients of the product.
14. Patient must not intend to use cannabinoids, cocaine, or nonprescribed opiates.
15. Involvement in the planning and/or conduct of the study (applies to both Noema staff and/or staff at the study site).
16. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
17. Previous randomization in the present study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald A Maguire, M.D., Principal Investigator — Clinical Innovations, Inc. dba CITrials (a CenExel company)
Locations (9):
- United States (6):
  - Noema Investigator site, Bellflower, California
  - Noema Investigator site, Jacksonville, Florida
  - Noema Investigator site, Orlando, Florida
  - Noema Investigator site, Overland Park, Kansas
  - Noema Investigator site, Berlin, New Jersey
  - Noema Investigator site, Memphis, Tennessee
- Australia (3):
  - Noema Investigator site, Brookvale, New South Wales
  - Noema Investigator site, Miranda, New South Wales
  - Noema Investigator site, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants were not randomized due to withdrawal by patient (n=3), non-compliance with study drug (n=1) or physician decision (n=1), 3 were not eligible for randomization.
Period: Overall Study
Arm/Group | Active | Placebo
Started | 34 | 31
Full analysis set | 33 | 29
Completed | 19 | 26
Not Completed | 15 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (10.09) | 34.3 (10.25) | 32.6 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 31 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 9 | 19
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 0 | 1 | 1
Maguire-Leal-Garibaldi Self-rated Stuttering Scale [Mean (Standard Deviation); unit: score on a scale] | 32.1 (14.23) | 33.3 (11.16) | 32.7 (12.86)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of 6 Weeks in Total MLGSSS
Description: MLGSSS refers to Maguire-Leal-Garibaldi Self-rated Stuttering Scale. The scale includes ten questions that are assessed on a 0 to 10 scale with 0 being no impact and 10 being highest impact. The total score ranges from 0 to 100 with the higher the score the worse the stuttering.
Time Frame: 43 days
Population: The full analysis set was used to assess the outcome. The full analysis set includes patients randomized who had at least one dose of study treatment and post randomization MLGSSS assessed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 33 | 29
Score on a scale | -7.0 (13.32) | -5.5 (6.72)

2. Secondary Outcome: Change From Baseline in Sheehan Disability Scale
Description: The Sheehan Disability Scale (SDS) is a brief, self-report tool that assesses disability or functional impairment in the domains of (1) Work/School life, (2) Social life, and (3) Family life/home responsibilities. Each is assessed on a 10 point scale with 0 being no impact, and 10 being highest impact. Each item is rated from 0 (not at all) to 10 (extremely) impairment. Each domain score is added to provide a total score from 0-30 total score with 0 (no impairment) and 30 is severe impairment. The change from the Baseline assessment have been provided.
Time Frame: Up to 71 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 33 | 29
score on a scale | -0.6 (8.23) | -1.3 (5.82)

3. Secondary Outcome: Change From Baseline to End Point in Clinician-rated Stuttering Severity Instrument-4
Description: SSI-4 is a validated scale to evaluate speech fluency including frequency, duration, physical concomitants and the naturalness of the speech. The score ranges from 10 (mildest) to 46 (most severe). The results show the change from Baseline in the SSI-4
Time Frame: Up to 71 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 33 | 29
units on a scale | -3.0 (6.5) | -2.7 (4.78)

4. Post Hoc Outcome: Change in MLGSSS From Baseline in More Severe Population
Description: MLGSSS refers to Maguire-Leal-Garibaldi Self-rated Stuttering Scale. The scale includes ten questions that are assessed on a 0 to 10 scale with 0 being no impact and 10 being highest impact. The total score ranges from 0 to 100 with the higher the score the worse the stuttering. Analysis of a subset of participant with a Baseline MLGSSS of > 24, in other words this analysis excludes those with mild stuttering as measured by MLGSSS. See the description for the first outcome measure for a description of the scale. The results show the change from baseline.
Time Frame: Up to 71 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale | -14.8 (12.54) | -9.1 (8.81)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial (71 days)
Groups:
- Active: Escalating doses of NOE-105 capsules
  NOE-105: Escalating dose levels of NOE-105 will be given and maximum tolerated dose will be maintained. The adverse event rates could not be allocated per dose because the dose titration occurred over a period of 4 weeks or util maximum tolerated dose reached. Down titration was also allowed
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 23/34 | 13/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=34) | Placebo (N=31)
Sedation (Nervous system disorders) | 8 | 1
Dystonia (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 2 | 1
Bradykinesia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Akathisia (Nervous system disorders) | 3 | 0
Restlessness (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Apathy (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Eye infection and bacterial (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Dysphemia (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT05583955/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT05583955/SAP_001.pdf